CLINICAL TRIAL: NCT01156532
Title: Observational Study; Clinical Effectiveness and Impact on Health-related Quality of Life in Peruvian Patients With Psoriasis After 16 Weeks of Adalimumab Therapy
Brief Title: Clinical Effectiveness and Impact on Health-related Quality of Life in Peruvian Patients With Psoriasis After 16 Weeks of Adalimumab Therapy
Status: Terminated | Type: Observational
Why Stopped: This study was prematurely terminated due to low enrollment and not for safety reasons.
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-261
Record Dates: First submitted 2010-07-01; First posted 2010-07-05 (Estimated); Results first posted 2014-08-25 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Moderate to Severe Psoriasis
Keywords: adalimumab therapy; Psoriasis; observational study
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Adalimumab Treatment in Participants with Psoriasis: Participants with moderate to severe chronic plaque psoriasis defined as Psoriasis Area and Severity Index (PASI) ≥ 10 and body surface area ≥ 10% with or without psoriatic arthritis, who have an adalimumab therapy indication because they are candidates for systemic therapy or phototherapy and other systemic therapies are medically less appropriate.

SUMMARY:
Adalimumab has recently been authorized for active psoriasis in Peru and local experience is very low. The aim of this study is to obtain Peruvian data of clinical effectiveness and impact on health-related quality of life with the use of adalimumab in participants with chronic plaque psoriasis complying with the dosing and monitoring recommendations of the local approved label.

ELIGIBILITY:
Inclusion Criteria:

* Participants with moderate to severe chronic plaque psoriasis defined as Psoriasis Area and Severity Index (PASI) ≥ 10 and body surface area ≥ 10% with or without psoriatic arthritis, who have an adalimumab therapy indication because they are candidates for systemic therapy or phototherapy and other systemic therapies are medically less appropriate
* Participant is capable of and willing to give written informed consent and to comply with the requirements of the study protocol

Exclusion Criteria:

* Participants should not be enrolled if they cannot be treated in accordance with the local product label
* Participants enrolled into another study or clinical trial
* History of hepatitis B infection
* History of neurologic symptoms suggestive of central nervous system demyelinating disease
* History of cancer or lymphoproliferative disease (other than successfully treated non-melanoma skin cancer or localized carcinoma in situ of the cervix)
* Active tuberculosis infection before initiating adalimumab treatment or latent tuberculosis infection not able to take complete prophylactic treatment
* Pregnant or lactating female, demonstrated by a pregnancy test before entering the study and willing to use a contraceptive method
* Use of another anti-tumoral necrosis factor previously
* History of congestive heart failure
* Any other condition that according to the criteria of the participating investigator represents an obstacle for study conduction and/or subjects participants to an unacceptable risk
* Participants with active infection including chronic or localized infections until infections are controlled
* History of sensitivity to latex
* Participants who will receive concomitant phototherapy and systemic therapy during adalimumab therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with moderate to severe psoriasis who receive adalimumab therapy according to standard clinical practice at Peruvian hospitals/clinics.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Uribe, MD, Study Director — AbbVie
Locations (3):
- Peru (3):
  - Site Reference ID/Investigator# 35783, Lima
  - Site Reference ID/Investigator# 56700, Lima
  - Site Reference ID/Investigator# 43147, Trujillo

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adalimumab Treatment in Participants With Psoriasis
Started | 30
Completed | 28
Not Completed | 2
Not completed — Family Reasons | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab Treatment in Participants With Psoriasis
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reaching a Psoriasis Area and Severity Index 75 (PASI-75) Response
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). PASI-75 responders are the participants who achieved at least a 75% reduction (improvement) from baseline in PASI score at Week 16. The mean PASI improvement was calculated using a linear regression model.
Time Frame: Baseline to Week 16
Population: Participants with available data. One participant was excluded from the analysis because only baseline and not follow-up information was available. Furthermore, 3 participants did not have their PASI measurement available either at baseline or at their last follow-up visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab Treatment in Participants With Psoriasis
Number analyzed (Participants) | 26
percentage of participants | 78 [61 to 95]

2. Primary Outcome: Percentage of Participants Reaching a Minimal Important Difference (MID) in the Dermatology Life Quality Index (DLQI) Score
Description: Dermatology Life Quality Index (DLQI) score is a participant-reported outcome consisting of a set of 10 questions regarding the degree to which the participant's skin has affected certain behaviors and quality of life over the last week. Responses to each are: very much (score of 3), a lot, a little, or not at all (score of 0). The DLQI score ranges from 0 (best) to 30 (worst); the higher the score, the more quality of life is impaired. MID for the DLQI was defined as a score decrease from baseline of 2.3 to 5. The mean DLQI improvement was calculated using a linear regression model.
Time Frame: Baseline to Week 16
Population: Participants with available data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab Treatment in Participants With Psoriasis
Number analyzed (Participants) | 26
percentage of participants | 92 [83 to 100]

3. Secondary Outcome: European Quality of Life 5 Dimensions (EQ-5D) Index Score at Baseline and Week 16
Description: EQ-5D is a self-reported health outcome which measures mobility, self-care, usual activities, pain discomfort, anxiety, and depression. An overall score is derived that measures from -0.59 (worst) to +1 (best). Improvement was defined as a mean score increase of at least 0.2.
Time Frame: Baseline, Week 16
Population: Participants with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab Treatment in Participants With Psoriasis
Number analyzed (Participants) | 26
units on a scale
  Baseline | 0.48 (0.40)
  Week 16 | 0.80 (0.32)

4. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An adverse event was considered an SAE if it met any of the following criteria: death of the participant; life-threatening event; hospitalization; prolongation of hospitalization; congenital anomaly; persistent or significant disability/incapacity; an important medical event requiring medical or surgical intervention to prevent serious outcome; spontaneous or elective abortion. SAEs included the occurrence of tuberculosis, opportunistic infection, and malignancy.
Time Frame: From the time of informed consent until 70 days (5 half-lives) after the last dose of study drug (treatment was 16 weeks).
Population: Participants who received at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Adalimumab Treatment in Participants With Psoriasis
Number analyzed (Participants) | 29
participants | 1

5. Secondary Outcome: Adherence to Adalimumab Treatment
Description: Adherence was measured by how many times a participant had a discontinuation (i.e., missed a study dose) during the 16 weeks of treatment.
Time Frame: up to 16 weeks
Population: Participants who received at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Adalimumab Treatment in Participants With Psoriasis
Number analyzed (Participants) | 29
participants
  No Missed Doses | 24
  One Missed Dose | 3
  Two Missed Doses | 2

6. Secondary Outcome: Mean Psoriasis Area and Severity Index (PASI) Score Over Time
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). The mean PASI improvement was calculated using a linear regression model.
Time Frame: Baseline, Week 4, Week 8, Week 16
Population: Participants with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab Treatment in Participants With Psoriasis
Number analyzed (Participants) | 26
units on a scale
  Baseline | 22.8 (9.0)
  Week 4 | 10.6 (9.8)
  Week 8 | 6.7 (8.4)
  Week 16 | 4.2 (9.1)

7. Secondary Outcome: Mean Dermatology Life Quality Index (DLQI) Score Over Time
Description: DLQI score is a participant-reported outcome consisting of a set of 10 questions regarding the degree to which the participant's skin has affected certain behaviors and quality of life over the last week. Responses to each are: very much (score of 3), a lot, a little, or not at all (score of 0). The DLQI score ranges from 0 (best) to 30 (worst); the higher the score, the more quality of life is impaired. The mean DLQI improvement was calculated using a linear regression model.
Time Frame: Baseline, Week 4, Week 8, Week 16
Population: Participants with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab Treatment in Participants With Psoriasis
Number analyzed (Participants) | 26
units on a scale
  Baseline | 20.3 (5.5)
  Week 4 | 10.8 (6.0)
  Week 8 | 5.9 (5.5)
  Week 16 | 4.6 (7.9)

ADVERSE EVENTS:
Time Frame: From the time of informed consent until 70 days (5 half-lives) after the last dose of study drug (treatment was 16 weeks).
Description: Adverse events are reported for all participants who received at least one dose of study treatment.
Arm/Group | Adalimumab Treatment in Participants With Psoriasis
Serious Adverse Events (participants affected / at risk) | 1/29
Other Adverse Events (participants affected / at risk) | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab Treatment in Participants With Psoriasis (N=29)
Cellulitis (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
Although a sample of 75 participants was originally planned, only 30 participants were enrolled in this study. The limited sample size can result in a potential sampling bias that cannot be tested.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.